CLINICAL TRIAL: NCT05640895
Title: The Effect of Entry Site Distance From Limbus on Perceived Pain During Intravitreal Injection of Anti-VEGF (Vascular Endothelial Growth Factor) Agents
Brief Title: Intravitreal Injection Site and Perceived Pain
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0228
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Pain
Keywords: Intravitreal injection; Retinal diseases; Age-related macular degeneration; Diabetic retinopathy; Retinal vein occlusion; Limbus; Quadrants (regions) of the eye; Injection site; Pseudophakic/aphakic eyes; Phakic eyes; Pars plana; Ciliary body; Vitrectomy; Crystalline lens; Retina; Bevacizumab; Ranibizumab; Aflibercept; Diabetic macular edema; Anti-VEGF (Vascular Endothelial Growth Factor); Vabysmo
MeSH Terms: conditions — Pain; Retinal Diseases; Macular Degeneration; Diabetic Retinopathy; Retinal Vein Occlusion; Aphakia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Intravitreal injection site — Intravitreal injections will be made at varying sites; patients will report on pain perception

SUMMARY:
The objective of this study is to explore the perception of pain during intravitreal injection related to the distance of the entry site from the limbus.

DETAILED DESCRIPTION:
In this pilot cross-over study, the investigators aim at exploring a factor not studied yet on the perception of pain during the injection procedure, and that is the distance of the entry site from the limbus.

Study population: Pseudophakic patients needing multiple intravitreal injections. In case of bilateral eligibility, one eye per patient will be included (randomly- based on a random chart).

Intervention: two injections per eye, will be included in the study. All steps of the technique will be similar between the two injections except for the entry site distance from the limbus, which will be 3.5 in one and 4.00 mm in the other. To prevent bias, the first injection entry distance will be randomly selected (based on a randomized chart).

The patient is blind to the entry distance, and a questionnaire with a visual analog pain scale will be given to the patient by a technician (to prevent any bias) to be filled after the injection. The analog pain scale is a scale of numbers from 0 to 10 representing the degree of patient's perceived pain. A score of 0 indicates no perception of pain; a score of 10 indicates a perception of the worst pain possible. The scale is also illustrated with face emojis corresponding to a written description of pain perception from no perception of pain, represented by a green, fully smiling face to perception of the worst pain possible, represented by a red, crying, fully frowning face.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -100 years
* Diagnosis of diabetic macular edema, age related macular degeneration, or retinal vein occlusion
* Treated with bevacizumab, ranibizumab, aflibercept
* The need for at least two intravitreal injections
* Pseudophakia

Exclusion Criteria:

* Texas Department of Corrections medical records
* Under 18 years-of-age
* First intravitreal injection experience of patient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be from university eye clinics scheduled to undergo intravitreal injections
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Visual scale analogues for pain | Immediately post-injection
  Self-reported perception of pain according to analogue pain scale. The analog pain scale is a scale of numbers from 0 to 10 representing the degree of patient's perceived pain. A score of 0 indicates no perception of pain; a score of 10 indicates a perception of the worst pain possible. The scale is also illustrated with face emojis corresponding to a written description of pain perception from no perception of pain, represented by a green, fully smiling face to perception of the worst pain possible, represented by a red, crying, fully frowning face.

CONTACTS AND LOCATIONS:
Overall Officials: Touka K Banaee, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Peyman GA, Lad EM, Moshfeghi DM. Intravitreal injection of therapeutic agents. Retina. 2009 Jul-Aug;29(7):875-912. doi: 10.1097/IAE.0b013e3181a94f01. PMID 19584648
- [Result] Gambrell J, Schaal S. Topical anesthesia for intravitreal injection. Expert Opin Drug Deliv. 2012 Jul;9(7):731-3. doi: 10.1517/17425247.2012.685156. Epub 2012 Jun 4. PMID 22657949
- [Result] Tewari A, Shah GK, Dhalla MS, Blinder KJ. Surface anesthesia for office-based retinal procedures. Retina. 2007 Jul-Aug;27(6):804-5. doi: 10.1097/IAE.0b013e31804b4081. No abstract available. PMID 17621193
- [Result] Karimi S, Mosavi SA, Jadidi K, Nikkhah H, Kheiri B. Which quadrant is less painful for intravitreal injection? A prospective study. Eye (Lond). 2019 Feb;33(2):304-312. doi: 10.1038/s41433-018-0208-y. Epub 2018 Sep 10. PMID 30202072